CLINICAL TRIAL: NCT05634239
Title: Senior Health Clinic for 75-year-old Home-dwelling Finns
Brief Title: Senior Health Clinic Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Marika Salminen, PhD, associate professor, University of Turku
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 87/1801/2019
Record Dates: First submitted 2022-11-21; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Cardiovascular Diseases; Dementia; Frailty
Keywords: Health Clinic; Prevention; Home-dwelling; Older people; Functional ability
MeSH Terms: conditions — Cardiovascular Diseases; Dementia; Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health check (Experimental)
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Health Education — Interview, clinical examination and health education conducted by the clinic nurse.
  Appointment with the physiotherapist including the assessment of physical functioning, use of assistive mobility devices, and amount of help needed in activities of daily living.

SUMMARY:
Turku Senior Health Clinic study The Turku Senior Health Clinic Study was targeted to 75-year-old citizens with an underlying idea that at that age it would be almost the last moment to nudge people towards healthy lifestyle and taking care of their health and functional ability to maintain independent living.

The short-term aims of the Turku Senior Health Clinic Study are to survey health and functional statuses and prevalence of specified risk factors for CVDs, dementia, frailty, and functional decline of 75-year-old independently home-dwelling citizens of the city of Turku. The aims also include assessment the frequency of follow-up treatments needed, and recommendations given for lifestyle changes and evidence-based drug treatment, as well as fulfillment of these recommendations. Also, participants feedback on the Turku Senior Health Clinic will be assessed. In addition, based on the results, recommendation for the content and implementation of preventive health clinic targeted to older people will be provided. The long-term aim of the research project is to assess the effects of the Turku Senior Health Clinic on the need of institutional care and home care as well as the cost-effectiveness of the clinic during the 10-year follow-up. For this purpose, participants of the Senior Health Clinic Study will be compared to that of non-participants and earlier cohorts of 75-year-olds in terms of the use of home care and institutional care.

ELIGIBILITY:
Inclusion Criteria:

* citizens of Turku
* home-dwelling

Exclusion Criteria:

* use of munical home care

Ages: 75 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Use of home care and institutional care. | 10 year
  Use of the municipal home care and institutional care among participant, non-participants and earlier cohorts from local registers.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Viikari, Study Director — University of Turku
Locations (1):
- University of Turku, Turku, University of Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salminen M, Luther-Tontasse E, Koskenniemi J, Vahlberg T, Wuorela M, Viitanen M, Korhonen P, Viikari L. Factors contributing to self-rated health in community-dwelling independent 75-year-old Finns: a population-based cross-sectional cohort study. BMC Geriatr. 2025 Mar 1;25(1):141. doi: 10.1186/s12877-025-05794-z. PMID 40025413
- [Derived] Salminen M, Stenholm S, Koskenniemi J, Korhonen P, Pitkanen T, Viikari P, Wuorela M, Viitanen M, Viikari L. Senior Health Clinic for 75-year-old home-dwelling Finns - study design, clinic protocol and non-response analysis. BMC Health Serv Res. 2023 Mar 2;23(1):210. doi: 10.1186/s12913-023-09199-9. PMID 36864394